CLINICAL TRIAL: NCT00623662
Title: Metabolic Preconditioning Using Intravenous Dextrose: a Novel Strategy to Improve Hepatic Function After Liver Resection
Brief Title: Preoperative Glucose Infusion: a Novel Strategy to Improve Liver Function After Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ralph Lattermann, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GEN-07-075; CIHR 183635
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Hepatic Insufficiency; Liver Failure
Keywords: Glucose infusion; Liver function; Liver resection; Albumin synthesis; Stable isotopes
MeSH Terms: conditions — Hepatic Insufficiency; Liver Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Glucose infusion.
  Interventions: Other: Preoperative glucose infusion
- 2 (Placebo Comparator): Normal saline infusion.
  Interventions: Other: Preoperative normal saline infusion

INTERVENTIONS:
Other: Preoperative glucose infusion — Glucose infusion from 15:00 on the day before the operation until beginning of surgery.
  Arms: 1
Other: Preoperative normal saline infusion — Normal saline infusion from 15:00 on the day before surgery until beginning of the operation.
  Arms: 2

SUMMARY:
The goal of the study is to determine whether intravenous glucose administration before liver resection preserves hepatic glycogen resulting in improved hepatic metabolic function after the operation.

We further investigate whether the benefit of avoiding preoperative fasting is more pronounced in patients undergoing more extensive liver resection.

DETAILED DESCRIPTION:
Background. With a reported incidence of up to 70%, liver failure is the most frequent complication necessitating intensive care and prolonging hospital stay. Animal studies suggest that the glycogen content of the liver is a key regulator of liver function and that glycogen depletion, a mandatory consequence of preoperative fasting, is associated with poor clinical outcome.

The results of a pilot study demonstrate that metabolic preconditioning, i.e. the avoidance of preoperative fasting by intravenous administration of dextrose preserves hepatic glycogen and prevents hepatic dysfunction after liver resection. Liver function in this protocol was assessed by a score originally proposed by Schindl including serum concentrations of total bilirubin and lactate, prothrombin time and degree of encephalopathy. Due to alterations induced by anesthesia and surgery, e.g. blood loss necessitating transfusion, hypothermia, inflammatory responses and use of drugs with impact on hepatobiliary metabolism, liver function scores do not necessarily reflect functional integrity and metabolic capacity of the liver. In contrast, measuring the production of proteins that are exclusively synthetized by hepatocytes such as albumin allows a more specific and quantitative assessment of hepatic performance under perioperative conditions.

Hypothesis. We propose a randomized double-blinded study to test the hypothesis that, in patients scheduled for resection of liver cancer, metabolic preconditioning with intravenous dextrose preserves hepatic glycogen resulting in improved hepatic metabolic function postoperatively. We further hypothesize that the benefit of avoiding preoperative fasting is more pronounced in patients undergoing more extensive liver resection. Hepatic synthetic capacity will be assessed by measuring albumin synthesis using a stable isotope tracer technique.

Research plan. In order to test the validity of our assumptions, we will perform studies in patients scheduled for minor (study I; one or two liver segments, n=30) or major (study II; three or more liver segments, n=20) liver resection. In a double blinded fashion patients will be randomly assigned to receive either intravenous dextrose at 2 mg/kg/min or saline from 15:00 on the day before the operation until surgical skin incision. Metabolic processes at the organ level (liver, muscle), i.e. fractional synthesis rates of albumin, hepatic acute phase proteins (transthyretin (=prealbumin), fibrinogen, total plasma proteins) and muscle protein will be determined one day before and one day after the operation using primed-continuous infusions of L-[2H5]phenylalanine. Stable isotopes (L-[1-13C]leucine, [6,6-2H2]glucose) will be applied to assess dynamic changes in whole body protein and glucose metabolism before and after surgery, i.e. protein breakdown, amino acid oxidation, protein synthesis, glucose production and glucose uptake.

Significance. The demonstration that the preconditioning with dextrose preserves metabolic performance of the liver would have important implications for the clinical management of surgical patients with liver cancer. If preoperative dextrose administration attenuates hepatic dysfunction after liver resection, it will provide these patients with a readily available, safe and inexpensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class ≤3
* liver resection (one or more liver segments) for primary or secondary malignancy
* ability to give informed consent

Exclusion Criteria:

* signs of severe malnutrition or obesity: body mass index (BMI) <20 or >30 kg.m-2, more than 10% involuntary body weight loss over the preceding six months, serum albumin <35 g.L-1
* chronic viral liver disease
* diabetes mellitus
* significant cardiorespiratory, renal and neurological disease
* musculoskeletal or neuromuscular disease
* severe anemia (hemoglobin <10 g.dL-1)
* history of severe sciatica or back surgery or other conditions which contraindicate the use of an epidural catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Rate of albumin synthesis | One day before and one day after surgery

SECONDARY OUTCOMES:
Transthyretin synthesis, fibrinogen synthesis, whole body glucose and protein kinetics | One day before and one day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Lattermann, MD PhD, Principal Investigator — Department of Anaesthesia, McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec, Canada